CLINICAL TRIAL: NCT02715609
Title: A Phase I/II Dose-escalation and Dose-expansion Study of Disulfiram/Copper With Concurrent Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Disulfiram/Copper With Concurrent Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201604115
Record Dates: First submitted 2016-03-09; First posted 2016-03-22 (Estimated); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Disulfiram; Gluconates; Copper; Surgical Procedures, Operative; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Disulfiram, Copper, Surgery, Radiation therapy, Temozolomide (dose escalation - dose level 2) (Experimental): * Disulfiram (DSF) dose level 2=250mg.
  * Preoperative DSF/Copper (CU) x 3 days (optional)
  * Surgery performed per routine clinical care.
  * After surgery, evaluation to confirm the final pathological diagnosis as GBM (if not the patient will not continue with the 2nd part of the study).
  * Radiation therapy (RT) 4-6 weeks following surgery at 60 Gy in 30 daily fractions.
  * Temozolomide (TMZ) from Day 1 of RT to the last day of RT at a daily oral dose for a maximum of 49 days as per standard clinical care.
  * DSF daily and Cu three times daily during chemoradiotherapy as per preoperative dose.
  * 4-6 weeks after completion of chemoradiotherapy, adjuvant TMZ may be administered for 6 cycles. TMZ on Days 1-5 of every 28-day cycle. Daily DSF of 500mg will be continued with adjuvant TMZ for up to 6 cycles.
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate; Procedure: Surgery; Radiation: Radiation; Drug: Temozolomide
- Disulfiram, Copper, Surgery, Radiation therapy, Temozolomide (dose escalation - dose level 3) (Experimental): * Disulfiram (DSF) dose level 3=375mg.
  * Preoperative DSF/Copper (CU) x 3 days (optional)
  * Surgery performed per routine clinical care.
  * After surgery, evaluation to confirm the final pathological diagnosis as GBM (if not the patient will not continue with the 2nd part of the study).
  * Radiation therapy (RT) 4-6 weeks following surgery at 60 Gy in 30 daily fractions.
  * Temozolomide (TMZ) from Day 1 of RT to the last day of RT at a daily oral dose for a maximum of 49 days as per standard clinical care.
  * DSF daily and Cu three times daily during chemoradiotherapy as per preoperative dose.
  * 4-6 weeks after completion of chemoradiotherapy, adjuvant TMZ may be administered for 6 cycles. TMZ on Days 1-5 of every 28-day cycle. Daily DSF of 500mg will be continued with adjuvant TMZ for up to 6 cycles.
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate; Procedure: Surgery; Radiation: Radiation; Drug: Temozolomide
- Disulfiram, Copper, Surgery, Radiation therapy, Temozolomide (dose expansion) (Experimental): * Surgery performed per routine clinical care.
  * Radiation therapy (RT) 4-6 weeks following surgery at 60 Gy in 30 daily fractions.
  * Temozolomide (TMZ) from Day 1 of RT to the last day of RT at a daily oral dose for a maximum of 49 days as per standard clinical care.
  * Disulfiram (DSF) daily (250 mg) and Copper (Cu) three times daily during chemoradiotherapy.
  * 4-6 weeks after completion of chemoradiotherapy, adjuvant TMZ may be administered for 6 cycles. TMZ on Days 1-5 of every 28-day cycle. Daily DSF of 500mg will be continued with adjuvant TMZ for up to 6 cycles.
  * If a patient develops recurrent tumor during follow-up and plans to undergo another resection, he/she may opt for an optional preoperative DSF study prior to salvage surgery.
  Interventions: Drug: Disulfiram; Drug: Copper Gluconate; Procedure: Surgery; Radiation: Radiation; Drug: Temozolomide

INTERVENTIONS:
Drug: Disulfiram
  Other Names: DSF; Antabuse®
Drug: Copper Gluconate
  Other Names: Copper; Cu
Procedure: Surgery
Radiation: Radiation
Drug: Temozolomide
  Other Names: Temodar®

SUMMARY:
The proposed phase I/II study of disulfiram (DSF) for patients with presumed glioblastoma multiforme (GBM) based on magnetic resonance imaging (MRI) or biopsy, including administration before surgery and during adjuvant chemoradiotherapy. Patients will be treated with 3 days of preoperative DSF/copper (Cu) prior to their surgery (or biopsy), which will be followed by collection of tumor samples during surgery for analysis of drug uptake. After the surgery, patients will receive standard radiation therapy (RT) and temozolomide (TMZ) with the addition of concurrent DSF/Cu.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GBM or its histological variants (WHO grade IV). Patients who are participating in the optional preoperative pharmacokinetic study, may have presumed GBM based on clinical/radiological findings. However, patient must have histologically confirmed GBM before continuing to receive DSF with concurrent RT/TMZ.
* Expansion Cohort: must have a diagnosis of GBM (or its histological variants) with IDH, BRAF, or NF1 mutations. Confirmation of these mutations may be either by immunohistochemistry or next-generation sequencing
* At least 18 years of age.
* Karnofsky performance status (KPS) of at least 60%
* For patients who will participate in the optional pre-operative DSF pharmacokinetic study, they should be eligible for surgical resection for which at least 0.2 cubic cm or approximately 200 mg of tumor will be removed in additional to tumor specimen required for pathology evaluation. Patients enrolled after undergoing surgical resection or biopsy with histologically confirmed GBM are not required to meet this point of inclusion.
* Eligible for and planning to receive standard fractionated RT with concurrent TMZ.
* Willing to remain abstinent from consuming alcohol while on DSF.
* Willing to defer definitive surgery for one week while taking DSF and Cu. Patients who declined the optional pre-operative pharmacokinetic study or enrolled after undergoing surgical resection or biopsy with histologically confirmed GBM are not required to meet this point of inclusion.
* Meets the following laboratory criteria:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin > 10.0 g/dL (transfusion and/or ESA allowed)
  * Total bilirubin ≤ 2x institutional upper limit of normal (ULN)
  * AST and ALT < 3 x ULN
  * Serum creatinine < 1.5 x ULN or creatinine clearance > 50 mL/min (by Cockcroft-Gault)
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to take oral medication.
* Able to understand and willing to sign an IRB-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

* Receipt of any other investigational agents within 14 days prior to study treatment
* Enrolled on another clinical trial testing a novel therapy or drug.
* History of allergic reaction to DSF or Cu.
* Treatment with the following medications are contraindicated with DSF when taken within 7 days prior to the first dose of DSF + Cu: metronidazole, isoniazid, dronabinol, carbocisteine, lopinavir, paraldehyde, ritonavir, sertaline, tindazole, tixanidine, atazanavir. (Note: the following medications are not contraindicated but should be cautioned if taking concurrently with DSF: warfarin, phenytoin, theophylline, chlorzoxazone, chlordiazepoxide, diazepam. If the patient is taking warfarin, INR should be monitored closely. If the patient has to remain on phenytoin, its serum concentration and response should be monitored closely.
* Active or severe hepatic, cardiovascular, or cerebrovascular disease, including myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* History of idiopathic seizure disorder, psychosis, or schizophrenia.
* History of Wilson's disease or family member with Wilson's disease.
* History of hemochromatosis or family member with hemochromatosis.
* Pregnant and breastfeeding women will be excluded because of the known teratogenic effect of RT and the unknown effect of TMZ and DSF on fetal development. Women of childbearing potential must have a negative pregnancy test within 14 days of initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Started | 9 | 10 | 16
Completed | 8 | 10 | 15
Not Completed | 1 | 0 | 1
Not completed — Patient only completed pre-operative treatment | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion) | Total
Number analyzed (Participants) | 9 | 10 | 16 | 35
Age, Continuous [Median (Full Range); unit: years] | 56 [22 to 72] | 48 [23 to 78] | 51.5 [29 to 73] | 51 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 3 | 14
  Male | 6 | 2 | 13 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 9 | 9 | 15 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of DSF (Dose-escalation Phase Only)
Description: * The maximum tolerated dose (MTD) of DSF is defined as the dose level at which 20% of the cohort experience dose-limiting toxicity (DLT) within 18 weeks from start of RT (or 12 weeks from the end of RT if there is a delay in RT). MTD is assessed from the first dose of DSF in combination with TMZ and RT; patients will not be assessed for DLT during the pre-surgery period when they are receiving the lead-in doses of DSF.
  * A DLT is defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications/TMZ which occurs within 18 weeks following the first dose of DSF with RT+TMZ (corresponding to approximately 6 weeks during RT and 12 weeks after RT)
Time Frame: Estimated to be 2 years and 28 weeks
Population: One participant was not evaluable in dose escalation - dose level 2 as the participant did not receive DSF + RT + TMZ. This outcome measure is not for dose expansion portion of the trial.
Measure: Number; unit: mg
Groups:
- Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2 & 3): * Disulfiram (DSF) dose level 2=250mg, dose level 3=375mg
  * Preoperative DSF/Copper (CU) x 3 days (optional)
  * Surgery performed per routine clinical care.
  * After surgery, evaluation to confirm the final pathological diagnosis as GBM (if not the patient will not continue with the 2nd part of the study).
  * Radiation therapy (RT) 4-6 weeks following surgery at 60 Gy in 30 daily fractions.
  * Temozolomide (TMZ) from Day 1 of RT to the last day of RT at a daily oral dose for a maximum of 49 days as per standard clinical care.
  * DSF daily and Cu three times daily during chemoradiotherapy as per preoperative dose.
  * 4-6 weeks after completion of chemoradiotherapy, adjuvant TMZ may be administered for 6 cycles. TMZ on Days 1-5 of every 28-day cycle. Daily DSF of 500mg will be continued with adjuvant TMZ for up to 6 cycles.
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2 & 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 18 | 0
mg | 375 |

2. Primary Outcome: Kaplan-Meier Estimate of Overall Survival (Dose-expansion Phase Only)
Time Frame: 1 year
Population: This outcome measure is for participants enrolled in dose expansion only.
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 0 | 0 | 15
percentage of participants-Kaplan Meier |  |  | 80

3. Primary Outcome: Kaplan-Meier Estimate of Overall Survival (Dose-expansion Phase Only)
Time Frame: 2 years
Population: This outcome measure is for participants enrolled in dose expansion only.
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 0 | 0 | 15
percentage of participants-Kaplan Meier |  |  | 67

4. Primary Outcome: Kaplan-Meier Estimate of Overall Survival (Dose-expansion Phase Only)
Time Frame: 3 years
Population: This outcome measure is for participants enrolled in dose expansion only.
Measure: Number; unit: percentage of participants-Kaplan Meier
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 0 | 0 | 15
percentage of participants-Kaplan Meier |  |  | 52

5. Primary Outcome: Mean Overall Survival (Dose-expansion Phase Only)
Time Frame: Through completion of follow-up (up to 5 years)
Population: This outcome measure is for participants enrolled in dose expansion only.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 0 | 0 | 15
months |  |  | 37.4 [26.2 to 48.6]

6. Secondary Outcome: Toxicity of DSF When Given Concurrently With Radiation Therapy and Temozolomide as Measured by the Grade and Frequency of Grade 2 or Greater Adverse Events Related to DSF
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: Through completion of DSF treatment (up to 38 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 8 | 10 | 15
Participants
  Grade 2 nausea | 0 | 2 | 2
  Grade 2 diarrhea | 0 | 1 | 0
  Grade 2 fatigue | 1 | 1 | 3
  Grade 3 fatigue | 0 | 1 | 0
  Grade 2 alanine aminotransferase increased | 1 | 0 | 0
  Grade 3 alanine aminotransferase increased | 0 | 1 | 2
  Grade 4 alanine aminotransferase increased | 0 | 1 | 0
  Grade 2 aspartate aminotransferase increased | 0 | 1 | 0
  Grade 3 aspartate aminotransferase increased | 0 | 1 | 2
  Grade 2 fall | 0 | 1 | 0
  Grade 2 ataxia | 1 | 0 | 0
  Grade 3 confusion | 0 | 1 | 0
  Grade 2 urinary incontinence | 1 | 1 | 0
  Grade 3 urinary incontinence | 0 | 0 | 1
  Grade 4 neutrophil count decreased | 0 | 0 | 1
  Grade 2 anorexia | 0 | 0 | 1
  Grade 2 dizziness | 0 | 0 | 1

7. Secondary Outcome: Intratumor and Plasma Concentration of DSF Metabolite (Ditiocarb-copper Complex)
Description: Will be determined using mass spectrometer
Time Frame: At the time of surgery (day 4)
Population: Only 3 patients had tumor resection after preoperative DSF/Cu administration.
Measure: Number; unit: ng/mL
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 2 | 1
ng/mL
  Plasma CuET concentration - patient #1: number analyzed (Participants) | 1 | 0
  Plasma CuET concentration - patient #1 | 0.11 |
  Plasma CuET concentration - patient #2: number analyzed (Participants) | 0 | 1
  Plasma CuET concentration - patient #2 |  | 0.44
  Plasma CuET concentration - patient #3: number analyzed (Participants) | 1 | 0
  Plasma CuET concentration - patient #3 | 4.59 |
  Tumor CuET concentration - patient #1: number analyzed (Participants) | 1 | 0
  Tumor CuET concentration - patient #1 | 0.00 |
  Tumor CuET concentration - patient #2: number analyzed (Participants) | 0 | 1
  Tumor CuET concentration - patient #2 |  | 0.00
  Tumor CuET concentration - patient #3: number analyzed (Participants) | 1 | 0
  Tumor CuET concentration - patient #3 | 0.00 |

8. Secondary Outcome: Mean Progression-free Survival (PFS)
Description: Will be determined from the first day of RT to the time of tumor progression or death, whichever occurs first. Tumor progression will be determined using the RANO criteria.
Time Frame: Through completion of follow-up (up to 5 years)
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
Number analyzed (Participants) | 8 | 10 | 15
months | 24.4 [12.9 to 35.8] | 32.3 [13.0 to 51.7] | 34.5 [22.0 to 46.9]

9. Other Pre Specified Outcome: Rate of Pseudo-progression (PsP)
Description: -Pseudoprogression is defined as a transient increase of tumor after chemoradiotherapy that subsequently stabilizes without a change of therapy
Time Frame: Through completion of follow-up (up to 5 years)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Pharmacodynamic Studies on Glutamate Metabolism as Measured by Measurement of Glutamine Levels in Plasma and Tumor Tissues
Time Frame: Week 6
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pharmacodynamic Studies on Glutamate Metabolism as Measured by Measurement of Glutamate Levels in Plasma and Tumor Tissues
Time Frame: Week 6
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Time to Tumor Progression (TTP) (Dose-escalation Phase Only)
Description: -≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids. The absolute increase in any dimension must be at least 5mm when calculating the products
  * Significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy not caused by comorbid events
  * Any new measureable lesion
  * Clear clinical deterioration not attributable to other causes apart from the tumor (e.g. seizures, medication adverse effects, complications of therapy, cerebrovascular events, infection, and so on) or changes in corticosteroid dose
  * Failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease
Time Frame: Through completion of follow-up (up to 5 years)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pharmacodynamic Studies on Glutamate Metabolism as Measured by Measurement of Aspartate Levels in Plasma and Tumor Tissues
Time Frame: Week 6
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Pharmacodynamic Studies on Glutamate Metabolism as Measured by Measurement of Glucose Levels in Plasma and Tumor Tissues
Time Frame: Week 6
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Pharmacodynamic Studies on Glutamate Metabolism as Measured by Measurement of Lactate Levels in Plasma and Tumor Tissues
Time Frame: Week 6
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until the last dose of DSF (median length of follow-up 131 days, full range 2-288 days). All-cause mortality was collected from start of treatment through completion of follow-up (up to 5 years).
Arm/Group | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion)
All-Cause Mortality (participants affected / at risk) | 5/9 | 5/10 | 9/16
Serious Adverse Events (participants affected / at risk) | 3/9 | 5/10 | 7/16
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) (N=9) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) (N=10) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion) (N=16)
Death NOS (General disorders) | 0 | 0 | 4
Fever (General disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 2) (N=9) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Escalation - Dose Level 3) (N=10) | Disulfiram, Copper, Surgery, Radiation Therapy, Temozolomide (Dose Expansion) (N=16)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Elevated heart rate (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0
Diminished peripheral vision - left side (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Right peripheral field cut (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 4
Dental abscess (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 4 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1 | 1
Chills (General disorders) | 2 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0
Edema hands (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 8 | 7 | 11
Fever (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 2
Infusion related reaction (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 1
Cold (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Yeast infection (Infections and infestations) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 6 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 5 | 2 | 0
Weight loss (Investigations) | 2 | 0 | 0
White blood cell decreased (Investigations) | 2 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 1
Diabetes mellitus-steroid induced (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 2 | 3 | 5
Cognitive disturbance - aphasia (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 8 | 2 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 0
Dysphasia (Nervous system disorders) | 1 | 2 | 2
Facial muscle weakness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 6 | 3
Impaired balance (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Lightheadedness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 6 | 2 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 3
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 5 | 4 | 0
Tunnel vision (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 1
Confusion (Psychiatric disorders) | 3 | 3 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 5 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 3 | 1
Irritability (Psychiatric disorders) | 2 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
Dribbling with urination (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 2 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT02715609/Prot_SAP_000.pdf